CLINICAL TRIAL: NCT06388486
Title: Cytokine-Induced Transcription in Depressed Inpatients Undergoing Psychotherapy
Acronym: CitDip
Status: Completed | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Prof. Thomas Meyer, Clinical Professor, Head of the Molecular Psychocardiology laboratory, University Medical Center Goettingen
Other Study IDs: UMCGoettingen9/9/16
Record Dates: First submitted 2024-04-23; First posted 2024-04-29 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Psychotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Psychotherapy — Subject receive psychotherapy during hospital treatment.

SUMMARY:
The goal of this observational study is to measure the levels of cytokine-induced transcription factor activation in a cohort of depressed inpatients undergoing psychotherapy. The study aims to answer the following main questions:

* Do psychological traits (i.e.: social inhibition, negative affectivity, ...) affect the activation of immunomodulatory transcription factors (STAT3, NFkB) in depressed patients?
* Are subjects with these psychological traits affected differently by psychotherapeutic intervention?

Study subjects are assessed for their psychological and behavioral traits and receive psychotherapeutic care over several weeks during hospital treatment. Peripheral blood mononuclear cells are isolated from the study subjects, and activation of transcription factors is measured by flow cytometry.

DETAILED DESCRIPTION:
Study subjects are assessed for their psychological and behavioral traits and receive psychotherapeutic care over several weeks during hospital treatment. Peripheral blood mononuclear cells are isolated from the study subjects, and activation of transcription factors is measured by flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of current depression

Exclusion Criteria:

* inadequate knowledge of the German language
* unable to give informed consent
* severe psychiatric comorbidities, such as drug abuse and psychotic diseases
* deemed critically unstable by their treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Depressed inpatients, admitted for multimodal treatment, including psychotherapy.
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Change in depression | 6 weeks
  Hospital Depression and Anxiety Scale (HADS). The HADS instrument is a 14-item scale, with seven items relating to anxiety and seven relating to depression item. Each item on qestionnaire is scored from 0-3 resulting in a score between 0 and 21 for either anxiety or depression with higher scores meaning a worse outcome.

IPD SHARING:
Plan to Share IPD: No